CLINICAL TRIAL: NCT02371720
Title: Patient Centered Comprehensive Medication Adherence Management System to Improve Effectiveness of Disease Modifying Therapy With Hydroxyurea in Patients With Sickle Cell Disease
Brief Title: Patient Centered Comprehensive Medication Adherence Management System in Patients With Sickle Cell Disease
Acronym: SCD Mobile Dot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Lakshmanan Krishnamurti, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00074105
Record Dates: First submitted 2015-02-19; First posted 2015-02-26 (Estimated); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Adults - Mobile DOT (Experimental): Subjects with SCD that are older than 21 years old will receive comprehensive medication adherence management (Mobile DOT) after 1 month assessment period. The subjects will receive the Mobile DOT intervention for 24 months.
  Interventions: Behavioral: Mobile DOT
- Adults - standard of care then Mobile DOT (Active Comparator): Subjects with SCD that are older than 21 years old will receive standard of care for the first 12 months. They will then crossover to the comprehensive medication adherence management plan (Mobile DOT) after 1 month assessment period for the remaining 12 months.
  Interventions: Behavioral: Mobile DOT
- Children - Mobile DOT (Experimental): Subjects with SCD that are younger than 21 years old will receive comprehensive medication adherence management (Mobile DOT) after 1 month assessment period. The subjects will receive the Mobile DOT intervention for 24 months.
  Interventions: Behavioral: Mobile DOT
- Children - standard of care then Mobile DOT (Active Comparator): Subjects with SCD that are younger than 21 years old will receive standard of care for the first 12 months. They will then crossover to the comprehensive medication adherence management plan (Mobile DOT) after 1 month assessment period for the remaining 12 months.
  Interventions: Behavioral: Mobile DOT

INTERVENTIONS:
Behavioral: Mobile DOT — Daily reminders via text or email to send a video of themselves taking their Hydroxyurea, positive feedback, and be encouraged to contact the research coordinator with any questions, concerns, etc.
  Other Names: Comprehensive medication adherence management

SUMMARY:
The purpose of this research study is to learn about ways to help children and adults with sickle cell disease who are taking the medication, hydroxyurea.

DETAILED DESCRIPTION:
Sickle cell disease (SCD) is an inherited chronic multi-organ system disorder that affects approximately 100,000 individuals in the United States, mostly belonging to minority, under-served populations. SCD is associated with substantial morbidity, premature mortality, individual suffering, health care costs and loss of productivity. Hydroxyurea (HU) the only disease modifying therapy for SCD is efficacious in reducing complications such as pain crisis and acute chest syndrome and improving survival. It is however, vastly underutilized and poorly adhered to because of barriers at the health care system, provider, treatment, socioeconomic, and patient levels. The investigator's overarching hypothesis is that barriers to acceptance and adherence to HU are multi-factorial and that a structured set of interventions can lead to improved adherence to medication and patient centered outcomes.

ELIGIBILITY:
Inclusion Criteria:

* be >2 years of age up to 65 years of age, inclusive
* have a diagnosis of SCD, with either βS/βS, βS/βC, βS/βD, βS/β0, βS/βO-Arab, or βS/β+ genotype
* prescribed Hydroxyurea for at least the 6 months prior to study entry
* have daily access to a smart phone, tablet, personal computer or other device capable of producing and transmitting videos over the internet
* be willing and able to record and transmit videos

Exclusion Criteria:

* patient or caregiver refuses to take Hydroxyurea as treatment for SCD
* diagnosis of significant psychiatric disorder of the subject that could seriously impede the ability to participate in the study
* an assessment by the investigator that the subject will not comply with the study procedures outlined in the study protocol
* patients receiving automatic home delivery of medications since medication possession ratio is reflective of the patient initiation the refill when they have exhausted the home supply of HU

Ages: 2 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2014-06-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Medication Possession Ratio (MPR) | 12 months
  Proportion of days the patient is in possession of the medication in the study period

SECONDARY OUTCOMES:
Change in Hemoglobin (Hb) levels | Baseline, 24 months
  Change in hemoglobin levels from baseline to 24 months will be measured using the HemoCue® rapid test.
Change in mean cell volume (MCV) | Baseline, 24 months
  Change from baseline in MCV will be calculated as the value at 24 months minus the value at baseline. MCV is the average size of the red blood cells expressed in femtoliters. MCV is calculated by dividing the hematocrit (as percent) by the red blood cell (RBC) count in millions per microliter of blood, then multiplying by 10.
Change in fetal hemoglobin (HbF) levels | Baseline, 24 months
  Change from baseline in HbF will be calculated as the value at 24 months minus the value at baseline. HbF is expressed as a percentage.
Impact of adherence on clinical outcomes and healthcare utilization | Baseline, 24 months
  Health care utilization in the emergency department and hospitalization due to sickle cell related complications such as vaso-occlusive crisis (VOC) or acute chest syndrome (ACS). Retrospective chart review at baseline will be conducted to determine healthcare utilization.
Impact of adherence on patients' lives | Baseline, 24 months
  Impact of adherence on patients' lives measured using patient reported outcomes (PROMIS), surveys of school attendance, work absenteeism, out-of-pocket costs incurred by patients and their caregivers
Change in adherence with using Mobile-DOT | Baseline, 24 months
  Retrospective chart review at baseline will be conducted to determine medication possession rate (MPR) and then compared to the MPR at 24 months.
Acceptability of intervention and of Hydroxyurea | Baseline, 24 months
  Acceptability will be measured by Treatment Satisfaction Questionnaire for Medication-9 (TSQM-9) The TSQM is a 14-item subject-assessed evaluation of treatment medication including 4 factors, Effectiveness, Side Effects, Convenience, and Global Satisfaction, and it utilizes the following responses on a 7-point Likert scale: 1=Extremely Dissatisfied, 2=Very Dissatisfied, 3=Somewhat Dissatisfied, 4=Neither Satisfied Nor Dissatisfied, 5=Somewhat Satisfied, 6=Very Satisfied, 7=Extremely Satisfied. Scores range from 0-100, with 0 as extremely dissatisfied and 100 as extremely satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Lakshmanan Krishnamurti, MD, Study Chair — Emory University/Children's Healthcare of Atlanta
Locations (4):
- United States (4):
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - University of Illinois at Chicago, Chicago, Illinois
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania